CLINICAL TRIAL: NCT03978546
Title: Diagnostic Performance of Smart Supra Perimetry (SSP) in Comparison With Standard Automated Perimetry (SAP) and Ocular Coherence Tomography (OCT).
Brief Title: Diagnostic Performance of Smart Supra Perimetry (The DPSSP Study)
Acronym: DPSSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: University of Manchester (Other); Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 250459
Record Dates: First submitted 2019-05-16; First posted 2019-06-07 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Glaucoma, Suspect; Glaucoma
Keywords: glaucoma
MeSH Terms: conditions — Ocular Hypertension; Glaucoma | interventions — Tomography, Optical Coherence; Radionuclide Imaging

STUDY DESIGN:
Intervention Model Description: All participants will have the same examinations but in a randomised order, these examinations are: Humphrey Visual Fields Test (10-2 and 24-2, SITA Standard), OCT Scan (Cube scan, Wide angle and macula scan) and Smart Perimetry - Henson 9000.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-Glaucoma Patient Arm (Experimental): All participants will complete the same assessments
  Interventions: Diagnostic Test: Humphrey Visual Field Test; Diagnostic Test: Optical Coherence Tomography (OCT) Scan; Diagnostic Test: Smart Perimetry - Henson 9000
- Glaucoma Patient Arm (Experimental): All participants will complete the same assessments
  Interventions: Diagnostic Test: Humphrey Visual Field Test; Diagnostic Test: Optical Coherence Tomography (OCT) Scan; Diagnostic Test: Smart Perimetry - Henson 9000

INTERVENTIONS:
Diagnostic Test: Humphrey Visual Field Test — SITA Standard and 24-2 and 10-2 visual field tests
Diagnostic Test: Optical Coherence Tomography (OCT) Scan — Circle and Wide Angle Scans
Diagnostic Test: Smart Perimetry - Henson 9000 — 24+10-2 Smart Supra test

SUMMARY:
Early glaucomatous visual field changes can be missed with the routinely used Standard Automated Perimetry (SAP) and the 24-2 test pattern due to limited sampling of the central 10 degrees. While this shortcoming can be overcome with the addition of a 10-2 test, performing both tests places extra demand on the perimetric services (doubling test times) and patients.

Smart Supra Perimetry (SSP) uses a new faster algorithm that can complete both 24-2 and 10-2 test patterns in a similar time frame to a single 24-2 SAP test. This comparative study aims to determine the sensitivity and specificity (i.e. diagnostic accuracy) of SSP in identifying early glaucomatous visual field loss. A sample of 100 patients with early/suspect glaucoma will undergo SAP 24-2 and 10-2 (SITA algorithm) using Humphrey visual field perimetry and SSP 24+10-2 using Henson 9000. Eyes will be categorised into 2 groups i.e., glaucoma and non-glaucoma, on the basis of structural changes to the disc as evaluated by the clinician. The sensitivity and specificity of the SAP and SSP tests will be established along with test duration. The size and location of defects established with both the SAP and SSP strategies will also be compared.

ELIGIBILITY:
Inclusion Criteria:

* Reliable SAP visual field results (fixation loss < 33%, false positive < 15% and false negative < 20%).
* Visual acuity better or equal to 0.20 logMAR.
* Spherical refractive error within -6.00 to +6.00D and cylindrical error <2.00D
* No ocular co-morbidity likely to affect the visual field or OCT results.
* Age: 40-80 yrs

Additional inclusion criteria for glaucomatous group:

* Optic disc showing glaucomatous changes.
* SAP MD not worse than -6dB

Additional inclusion criteria non-glaucoma group:

* Normal SAP visual field data (MD, PSD, GHT within normal range)
* No evidence of glaucoma or other Ocular co-morbidity in the eye suitable for the study.

Exclusion Criteria:

Exclusion criteria glaucomatous and control groups:

• Anomalous discs, Tilted discs, myopic discs.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance of smart supra perimetry | 12 months
  Area under the curve for Smart Suprathrold Perimetry using probability thresholds to differentiate early glaucoma from non-glaucomatous visual fields.

SECONDARY OUTCOMES:
Diagnostic performance of Optical Coherent Tomography | 12 months
  Sensitivity and specificity for Optical Coherent Tomography in the detection of early glaucoma.
Diagnostic performance of Standard Automated perimetry | 12 months
  Sensitivity and specificity for Standard Automated perimetry in the detection of early glaucoma.

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester Royal Eye Hospital, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sukumar S, Harper RA, Tsamis E, Hood D, Henson DB. Diagnostic Accuracy of Smart Supra Perimetry in Comparison With Standard Automated Perimetry in the Detection of Early Glaucoma. J Glaucoma. 2025 Sep 1;34(9):710-718. doi: 10.1097/IJG.0000000000002596. Epub 2025 May 14. PMID 40366217